CLINICAL TRIAL: NCT00328848
Title: After Discharge Management of Low Income Frail Elderly (AD-LIFE)
Brief Title: After Discharge Management of Low Income Frail Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Summa Health System (Other)
Responsible Party: Principal Investigator, Susan E. Hazelett, Investigator, Summa Health System
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01HS014539-01A1 (AHRQ); 1R01HS014539-01A1 (AHRQ)
Record Dates: First submitted 2006-05-18; First posted 2006-05-22 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Heart Failure, Congestive; Coronary Arteriosclerosis; Atrial Fibrillation; Cerebrovascular Accident; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus; Hypertension; Osteoarthritis; Osteoporosis
Keywords: patient care management; chronic disease
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease; Atrial Fibrillation; Stroke; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus; Hypertension; Osteoarthritis; Osteoporosis; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention care management (Experimental): post dischsrge care management by a nurse care manager who performs in-home vistis and reports to a interdisciplinary team. Team generates care recommendations based on patient goals. PCP and care manager implement the care plan that is based on patient goals. Includes education, behavioral interventions, and coaching.
  Interventions: Behavioral: Behavioral

INTERVENTIONS:
Behavioral: Behavioral — Group Treatment(patient education, self management support, caregiver support)
Behavioral: behavioral — patient education, self management support, caregiver support

SUMMARY:
The purpose of this study is to determine whether comprehensive post-hospitalization interdisciplinary care management can be an effective care delivery model to improve outcomes in low-income frail elderly.

DETAILED DESCRIPTION:
This randomized trial will test the effectiveness of improved clinical practice through comprehensive care management in elderly patients with chronic illness and functional impairment discharged from an acute care hospital. For the intervention group, patient care will be coordinated by a nurse care manager who will perform a comprehensive in home assessment and provide patient education and self management support. The care manager will work with an interdisciplinary team (IT) to develop and implement a plan of care. Evidence based care plans will be implemented in collaboration with the patient, the primary care physician (PCP), the local Area Agency on Aging (AAoA), and other community social agencies. The care manager will provide frequent patient follow up across all providers to ensure integration of medical and social issues. Control patients will be referred to the local AAoA with no IT follow up. Although control patients will receive, through the AAoA, referrals for care and psychosocial support, the absence of a care manager and IT will, we expect, result in functional decline, lower quality of life, and higher health care costs.

The intervention (n=265) and control (n=265) groups will be compared at 1 year on a profile of health and well being using a multiple endpoint global hypothesis testing strategy. The global measure will be comprised of the following 5 domains: function, institutionalization, quality of life, quality of medical management, and quality of self management. Priority populations identified by AHRQ who are targeted in this study include the elderly, patients with chronic illnesses, low income (dual eligible), and patients with disabilities. This study also includes minorities, women, and patients who live in the inner city. Future economic analyses of benefits (for which alternative funding is currently being sought) will inform policy makers about funding care management in AHRQ priority populations.

ELIGIBILITY:
Inclusion Criteria:

* > 65 years old
* Confirmed or probable dual eligible
* Have at least one chronic illness (chronic obstructive pulmonary disease [COPD], diabetes, stroke/atrial fibrillation, ischemic heart disease, hypertension, congestive heart failure [CHF], osteoporosis, osteoarthritis) and at least 1 impaired activity of daily living (ADL) 11 or 2 impaired instrumental activities of daily living (IADLs)
* Be discharged home or to a skilled nursing facility (or acute rehabilitation) for a maximum of 8 weeks before being discharged to home

Exclusion Criteria:

* Enrolled in this health system's care management program
* Chemically dependent
* Those with a Mental Status Questionnaire score > 5
* Diagnosed psychosis
* Dialysis
* Terminal diagnosis/hospice

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 530 (Actual)
Dates: Start 2005-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Function | Length of Study
Quality of life | Duration
Quality of medical management | Duration

SECONDARY OUTCOMES:
Mortality | Duration
Opportunity costs of caregiver time | Duration

CONTACTS AND LOCATIONS:
Overall Officials: Kyle R Allen, DO, Principal Investigator — Riverside Health System

REFERENCES:
- [Background] Allen KR, Hazelett SE, Jarjoura D, Wright K, Fosnight SM, Kropp DJ, Hua K, Pfister EW. The after discharge care management of low income frail elderly (AD-LIFE) randomized trial: theoretical framework and study design. Popul Health Manag. 2011 Jun;14(3):137-42. doi: 10.1089/pop.2010.0016. Epub 2011 Feb 15. PMID 21323461